CLINICAL TRIAL: NCT00485251
Title: Prospective Randomized Trial of Hand-assisted Laparoscopic Right Hemicolectomy vs Total Laparoscopic Right Hemicolectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pamela Youde Nethersole Eastern Hospital (Other)
Responsible Party: Department of Surgery, Pamela Youde Nethersole Eastern Hospital, Hong Kong, Department of Surgery, Pamela Youde Nethersole Eastern Hospital, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CShan
Record Dates: First submitted 2007-06-11; First posted 2007-06-12 (Estimated); Last update posted 2009-11-25 (Estimated); Status verified 2009-11

CONDITIONS: Operation Time; Pain Score; Recurrence; Survival
Keywords: operation time in minutes; pain score from 1-10; recurrence; survival
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): hand assisted right hemicolectomy
  Interventions: Procedure: hand-assisted laparoscopic right hemicolectomy; Procedure: hand-assisted right hemicolectomy
- 2 (Active Comparator): laparoscopic right hemicolectomy
  Interventions: Procedure: total laparoscopic right hemicolectomy; Procedure: laparoscopic right hemicolectomy

INTERVENTIONS:
Procedure: hand-assisted laparoscopic right hemicolectomy — using the lap disc that allows the insertion of single and into the abdomen for operation
  Arms: 1
Procedure: total laparoscopic right hemicolectomy — using laparoscopic instruments for mobilization and dissection inside the abdomen
  Arms: 2
Procedure: hand-assisted right hemicolectomy — hand-assisted right hemicolectomy
  Arms: 1
Procedure: laparoscopic right hemicolectomy — using laparoscopic instruments for mobilization and dissection inside the abdomen
  Arms: 2

SUMMARY:
The operation used for treating cancer in this location of the colon is called right hemicolectomy. Currently the investigators have two methods of minimal access approach to the abdominal cavity in order to complete this operation:

1. Total Laparoscopic right hemicolectomy The operation is completed by laparoscopic instruments using video laparoscopy. At the end of the procedure, a small wound was created for the delivery of bowel and extracorporeal anastomosis.
2. Hand-assisted laparoscopic right Hemicolectomy A 6.5cm incision is used to allow insertion of one of the surgeon's hands into the abdomen. The operation is completed by the surgeon's hand and laparoscopic instruments, using video laparoscopy.

These two operations are essentially identical except for the surgical access. Both total laparoscopic and Hand-assisted laparoscopic surgery has been practiced in the United States and Europe for over 10 years. Studies from the United State and Europe have demonstrated the safety and the benefits of both techniques in terms of pain and recovery. In order to find out which one is a better procedure, the investigators are carrying out a clinical trial to compare the two surgical options in their short-term and long term outcomes.

The results of this study may have an impact on the care of similar patients in the future.

DETAILED DESCRIPTION:
Under ALL circumstances, the principles in the Declaration of Helsinki MUST be complied

One of the colorectal specialists (Dr CC Chung, Dr KK Yau, Dr JCH Wong and Dr. HY S Cheung) in the colorectal team will be informed. Clear explanation of the diagnosis, natural history of the disease, different treatment options, their likely outcomes and potential complications will be given. If the patient opts for surgical treatment, he/ she will be invited to enter the study. Further explanation about the study will then be given. The patient information sheet will be given. The patient will then be allowed with all the time he/she needed for decision.

Randomization:

By drawing from concealed envelopes into either the "total lap" (Total laparoscopic right hemicolectomy) or the "hand-assisted" (Hand-assisted laparoscopic right hemicolectomy) groups

The Operation:

1. Patients were put on a liquid diet the day before operation. All received mechanical bowel preparation the night before surgery,
2. Prophylactic antibiotics with be given:

   Cefuroxime 1.5gm IVI Metronidazole 500mg IVI on induction
3. Operation should be performed by two of the following surgeons under general anaesthesia:

   Dr HYS Cheung Dr. JCH Wong Dr CC Chung Dr KK Yau
4. either Total laparoscopic right hemicolectomy or Hand-assisted right hemicolectomy will be performed according to the randomization.

Standardized post-operative care:

1. All patients would receive patient control analgesia (PCA) in the form of intravenous bolus morphine in the immediate postoperative period. The dosage and regimen were reviewed by the anaesthetists in-charge, who would stop the PCA according to their usual practice. Thereafter, Pethidine (1mg/kg) was given intramuscularly every 4 hours on demand. In addition, two tablets of dologesic were prescribed orally every 4 hours on demand;
2. Resume diet and off intravenous fluid as tolerated;
3. The pain score was recorded from postoperative day 1 to day 7
4. Date of ambulation, postoperative mortality and pathology were recorded.

Discharge Criteria:

1. Ambulatory (or resume the pre-operative motility status)
2. Free from any complications that required inpatient management
3. Had at least one bowel motion
4. Did not require parental analgesia

Follow Up Arrangement:

1. They were reviewed by clinical oncologists as outpatients, and adjuvant chemotherapy were selectively offered based on the final histological staging of the disease
2. All patients were followed up in the surgical clinic according to the structured proforma. They were followed up 4-monthly in the first 3 years, and 6-monthly thereafter. CEA would be taken at each visit. CXR and ultrasound abdomen would be analyzed annually. Surveillance colonoscopy would be analyzed every 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed to have operable carcinoma of caecum and ascending colon and hepatic flexure were potential candidates.

Exclusion Criteria:

* Patient who did not give informed consent;
* Patient who were considered unfit for operative treatment;
* Patient presented as acute surgical emergencies, including intestinal obstruction, peritonitis, or pericolic abscess, etc.;
* Patients with metastatic diseases on preoperative work up;
* Patient with synchronous tumours or polyps which necessitate extended or additional resection;
* Patients with tumour size larger than 6.5cm in any dimension on preoperative imaging or invasion to contiguous organs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-02; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
operation time | minutes

SECONDARY OUTCOMES:
pain score, recurrence | pain score during postoperative hospital stay, recurrence for 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Hester YS Cheung, FRACS, Principal Investigator — Department of Surgery, Pamela Youde Nethersole Eastern Hosptial, Hong Kong
Locations (1):
- Pamela Youde Nethersole Eastern Hosptial, Hong Kong, Hong Kong